CLINICAL TRIAL: NCT02784210
Title: The Effect of Corticosteroids on Inflammation at the Edge of Acute Multiple Sclerosis Plaques: An Investigator-Blinded Study
Brief Title: Effect of Corticosteroids on Inflammation at the Edge of Acute Multiple Sclerosis Plaques
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160114; 16-N-0114
Record Dates: First submitted 2016-05-26; First posted 2016-05-27 (Estimated); Last update posted 2025-09-24 (Actual); Status verified 2025-07-25

CONDITIONS: Multiple Sclerosis
Keywords: Centripetal Enhancement; MRI; 7 Tesla; Gadolinium; MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Methylprednisolone; Prednisone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone (Experimental): 3 day course of intravenous methylprednisolone 1000 mg/day
  Interventions: Drug: Methylprednisolone
- prednisone (Experimental): 3-day course of oral prednisone 1250 mg/day
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Methylprednisolone — 3 days of corticosteroids (intravenous methylprednisolone at 1000 mg/day
  Arms: Methylprednisolone
Drug: Prednisone — 3 days of corticosteroids (oral prednisone at 1250 mg/day
  Arms: prednisone

SUMMARY:
Background:

Multiple sclerosis (MS) affects the brain, spinal cord, and optic nerves. MS lesions can appear on the MRI (magnetic resonance imaging) scans in many ways. Sometimes they light up from the outer edge and fill inward. This is called ring enhancement. Researchers think this type of lesion may not heal as well as others. Corticosteroids are the standard treatment to reduce symptoms of MS relapse. But there is no standard treatment for people with enhancing MS lesions without signs of MS relapse. Researchers want to see if a short-term high-dose course of corticosteroids helps heal those lesions.

Objective:

To study the effects of short-term high-dose corticosteroids on ring-enhancing MS.

Eligibility:

Adults ages 18 and older who:

* Have MS and a rim-enhancing lesion on a prior brain MRI
* Are enrolled in another NINDS protocol

Design:

Participants will be screened under another protocol

Participants will be randomly assigned to get either no treatment or 3 days of treatment with a corticosteroid.

Participants will have:

* 1 baseline visit
* 3 days of high-dose steroids, intravenous or oral. If IV, participants will receive methylprednisolone by IV each day. Participants will also be prescribed medicine to protect their stomach.
* Follow-up visits will be at week 13 and week 25 after randomization to treatment or no treatment.

Visits include medical history and physical exam. Participants will have blood and urine tests. Participants will also have neurological exams and MRIs. Participants lie on a table that slides into a cylinder. They are in the scanner 1.5-2 hours. They get a dye through a catheter: A needle guides a thin plastic tube into an arm vein.

DETAILED DESCRIPTION:
Objectives:

The primary aim of this pilot study is to assess the effects of short-term, high-dose corticosteroid administration on the 12-week evolution of multiple sclerosis lesions with centripetal enhancement pattern on magnetic resonance imaging (MRI), in particular with respect to the development of a hypointense rim on 7-tesla phase images. In our prior work, the phase rim has been associated with persistent deleterious inflammation with poor repair and ongoing neurodegeneration within lesions.

Study population:

Up to 30 multiple sclerosis patients with asymptomatic contrast-enhancing lesions will be enrolled. Patients are randomly assigned to either 3 days of corticosteroids (intravenous methylprednisolone at 1000 mg/day or oral prednisone at 1250 mg/day) or to no treatment.

Design:

This is a single-site study.Patients undergo serial brain MRIs with gadolinium-based contrast agent on both 3- and 7-tesla scanners over an approximate 25-week period. 3-tesla scans are obtained at baseline and week 25. 7-tesla scans are obtained at baseline and at weeks 13 and 25. Participants with one or more centripetal/rim-enhancing lesions at the baseline scan are randomized and followed. Clinical evaluation and blood testing are performed at baseline and weeks 13 and 25.

Outcome measures:

The primary outcome measure is the presence or absence, on the week-13 7-tesla scan, of a hypointense phase rim in each of the lesions followed over time. Secondary outcome measures include the presence or absence of a hypointense phase rim at week 25, as well as the lesion volume and intralesional median R1 relaxation rate at weeks 13 and 25. From 3-tesla scans, we will measure the change in normalized intralesional proton density-weighted and T1-weighted signal, as well as the R1 relaxation rate, between baseline and week 25. We will also assess for the presence or absence of a hypointense phase at 3T. Additional exploratory outcome measures, including clinical and immunological assessments, will also be collected.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Multiple sclerosis, as defined by the 2017 Revised McDonald Criteria;
* Age 18 or older;
* Ability to provide informed consent;
* Able to participate in study procedures and provide high-quality clinical research and imaging data, based on limited artifacts on prior MRI scans and, when possible to determine;
* Presence of a gadolinium enhancing lesion on the screening (3T or 7T) brain MRI that demonstrates either centripetal/rim enhancement or a phase rim, or both;
* Simultaneously participates in another screening or natural history protocol within the NINDS Neuroimmunology Clinic at the time of study entry.
* Willing to use birth control if able to conceive a child

EXCLUSION CRITERIA:

* Medical contraindications for MRI (e.g., any non-organic implant or other device such as a cardiac pacemaker or infusion pump or other metallic implants, objects, or body piercings that are not MRI-compatible or cannot be removed);
* Psychological contraindications for MRI (e.g., claustrophobia), to be assessed at the time the medical history is collected;
* Treatment with systemic steroids in previous 30 days (non-systemic administration of steroids, such as topical or local injection, is acceptable);
* Experiencing new neurological symptoms, with onset in previous 2 weeks, attributable to MS relapse;
* Pregnancy or current breastfeeding;
* Screening labs, only if required per current NIH Clinical Center guidelines for kidney-function screening before gadolinium-based MRI contrast, demonstrating estimated glomerular filtration rate <60 mL/min;
* Known hypersensitivity to gadolinium-based contrast agents;
* Medical contraindications to corticosteroid administration (e.g., diabetes, gastric ulcer)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
the presence or absence of a hypointense phase rim around each lesion followed over time | at 13 weeks
  At week 13, the presence or absence of a hypointense phase rim around each lesion followed over time.

SECONDARY OUTCOMES:
The change in normalized intralesional proton density-weighted and T1-weighted signal, as well as the R1 relaxation rate, from 3T scan. | week 25
  From 3-tesla scans, we willmeasure the change in normalized intralesional proton density-weighted and T1-weighted signal, as wellas the R1 relaxation rate, between baseline and week 25.
The presence or absence of a 3T hypointense phase rim around each lesion | at week 25
  The presence or absence of a 3T hypointense phase rim around each lesion at week and 25
The presence or absence of a hypointense phase rim around each lesion followed over time. | at week 25
  At week 25, the presence or absence of a hypointense phase rim around each lesion followed over time.
Lesion volume and intralesional median R1 relaxation rate as determined from the 7T MP2RAGE scan, | at week 13 and 25
  Lesion volume and intralesional median R1 relaxation rate at weeks 13 and 25, as determined from the 7T MP2RAGE scan, comparing corticosteroid and no-treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Reich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that results in publication
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after publication
Access Criteria: Will be shared under tech transfer agreements

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-N-0114.html